CLINICAL TRIAL: NCT01794117
Title: A Phase 2 Study of Anakinra in Inflammatory Pustular Dermatoses: Evaluation of Therapeutic Efficacy and Validation of Pathogenic Mechanisms
Brief Title: Anakinra for Inflammatory Pustular Skin Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Edward Cowen, M.D., Principal Investigator, National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130071; 13-AR-0071
Record Dates: First submitted 2013-02-15; First posted 2013-02-18 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Sneddon-Wilkinson; Acrodermatitis Continua of Hallopeau; Pustular Psoriasis; Palmoplantar Pustulosis
Keywords: Anakinra; Pustular Psoriasis; Palmoplantar Pustulosis; DITRA; Subcorneal Pustular Dermatosis
MeSH Terms: conditions — Psoriasis; Skin Diseases, Vesiculobullous | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A/Anakinra 100 mg/day (Experimental): An initial dose of anakinra 100 mg/day will be administered daily via self-administered subcutaneous injection. If active disease persists at this dose, anakinra dose may be escalated up to 200 mg/day injected subcutaneously daily at week 4 and 300mg at week 8.
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — An initial dose of anakinra 100 mg/day will be administered daily via self-administered subcutaneous injection. If active disease persists at this dose, anakinra dose may be escalated up to 200 mg/day injected subcutaneously daily at week 4 and 300mg/day at week 8.
  Other Names: Kineret

SUMMARY:
Background:

* Inflammatory pustular skin diseases are a type of autoinflammatory disease in which the immune system attacks the bodys tissues. These diseases cause painful and itchy skin rashes, eye and mouth irritation, joint pain and fever. Several drugs for treating these diseases suppress the immune system. However, they can cause severe side effects when taken over a long period of time.
* Interleukin 1 (IL-1) is a small protein that may be important in causing the inflammation seen in pustular skin disease. Anakinra is a drug that works by blocking IL-1. It has been effective in treating some inflammatory conditions such as rheumatoid arthritis. However, anakinra has not been studied for use in patients with pustular skin disease. Researchers want to see whether anakinra will be effective in treating pustular skin disease.

Objectives:

- To see if anakinra can be used to treat inflammatory pustular skin disease.

Eligibility:

- Individuals at least 18 years of age who have inflammatory pustular skin disease.

Design:

* Participants will be screened with a physical exam and medical history. Their disease will be evaluated with blood tests, urine tests and imaging studies. Skin biopsies may also be collected.
* Participants will have an initial visit to receive the first dose of anakinra. They will be shown how to give themselves daily injections of anakinra.
* Participants will take anakinra for up to 12 weeks as long as there are no severe side effects. During this time, they will keep a study diary to record the severity of any rashes, pustules, itching, fevers, and skin or joint pain. They will bring this diary to their study visits.
* Participants will have study visits at weeks 4, 8 and 12. Treatment will be monitored at these visits with blood tests, urine tests and physical exams. Depending on the effects of the treatment, participants may have the dose of anakinra increased or decreased.
* Participants will have a final study visit 4 weeks after they stop taking anakinra.

DETAILED DESCRIPTION:
Background:

* Inflammatory disorders that present with neutrophilic pustular skin lesions, including generalized pustular psoriasis, are characterized by severe cutaneous manifestations, generalized inflammation and significant morbidity.
* Recent studies in patients with phenotypically similar pustular diseases have identified two monogenic forms of neutrophilic pustular psoriasis implicating interleukin (IL)-1 in disease pathogenesis.

  * Deficiency of the Interleukin 1 (IL-1) receptor antagonist (IL1RN, DIRA) is an autosomal recessive condition characterized by severe generalized pustular eruptions in the neonatal period, osteopenia, lytic bone lesions, joint pain, respiratory insufficiency, thrombosis, elevated acute phase reactants and significant mortality. Patients with this condition have responded rapidly to IL-1 receptor antagonist, anakinra.
  * Deficiency of IL-36 receptor antagonist (IL-36RN/IL1F5, DITRA) is an autosomal recessive condition with episodic widespread pustular skin lesions, fevers and systemic inflammation defined by marked leukocytosis and elevated c-reactive protein.
* Both IL1RN and IL36RN/IL1F5 are highly expressed in epidermal keratinocytes, suggesting a role for keratinocytes in initiating innate immunity-mediated inflammatory skin diseases, and ultimately manifesting in a pustular phenotype.
* Patients with inflammatory pustular diseases often respond poorly to conventional treatment with methotrexate, cyclosporine and anti- tumor necrosis factor (TNF) agents.
* Two recent case reports describe patients with pustular psoriasis unresponsive to TNF inhibition who responded to anti-IL-1 receptor therapy with anakinra. We hypothesize that monogenic and polygenic inflammatory pustular skin diseases share common pathogenic mechanisms mediated by IL-1.
* We propose a phase 2 study that will utilize a collaborative bench-to-bedside approach, applying targeted anti-IL-1 therapy, novel imaging modalities, and laboratory techniques including immunohistochemistry, gene expression and cytokine studies, and in vitro manipulations of skin to dissect and validate pathways in these complex diseases.

Objectives:

-To characterize the clinical efficacy, optimal dosing and safety of anakinra in patients with pustular dermatoses.

Eligibility:

* Age greater than or equal to 18 years.
* Active macroscopic noninfectious pustular skin lesions involving greater than or equal to 5% of the total body surface area, or palmoplantar involvement.
* Histopathologic confirmation of epidermal neutrophilic pustulosis.
* Patients must have maintained a stable dose of immunosuppressant therapy, retinoids or anti-neutrophil therapy for 2 weeks prior to study initiation with resultant stable or worsening skin disease.
* Use of biologic agents requires a washout period of at least 3 half-lives prior to study initiation.
* Patients must have organ and marrow function as defined below:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * creatinine within normal institutional limits OR creatinine clearance >60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

Design:

* A 16-week, open-label phase 2 study.
* Patients will initially receive treatment with anakinra 100 mg/day by self-administered subcutaneous injection.
* Disease response will be assessed every 4 weeks, and determination of dose escalation will be made based on clinical assessment. Dose escalation can increase up to 200 mg/day, and for patients >75 kg up to 300 mg/day at the end of week 8.
* If a response is achieved with anakinra, other immunosuppressants administered for the purpose of treatment of pustular skin disease may be tapered per physician discretion.
* Clinical assessment, and laboratory and subjective data will be collected in-person every 4 weeks to determine disease response. Telephone assessments will be performed weekly.
* Twenty-five evaluable patients will be enrolled onto this trial. The accrual ceiling for this study will be set to 30.

ELIGIBILITY:
* INCLUSION CRITERIA

1.1 Females and males, aged greater than or equal to 18.

1.2 Patients must demonstrate active noninfectious inflammatory pustular skin lesions resembling pustular psoriasis and involving greater than or equal to 5% total body surface area, or palmoplantar involvement. Conditions may include, but are not be limited to, pustular psoriasis, Sneddon-Wilkinson disease, subcorneal pustular dermatosis, reactive arthritis, palmoplantar pustulosis, acrodermatitis continua of Hallopeau and palmoplantar pustular psoriasis.

1.3 Patients must have histopathologic confirmation of epidermal neutrophilic pustular skin disease.

1.4 If taking immunosuppressants, retinoids or anti-neutrophil therapy, participants must maintain stable doses of these medications during the 2 weeks prior to study initiation.

1.5 Patients must have stable topical medication regimen for 2 weeks prior to study initiation.

1.6 Patients must have normal organ and marrow function as defined below:

leukocytes greater than or equal to 3,000/mcL

absolute neutrophil count greater than or equal to1,500/mcL

platelets greater than or equal to 100,000/mcL

creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.

1.7 Quantiferon tuberculosis (TB) Gold must be performed for screening for mycobacterium tuberculosis infection. However, a tuberculin skin test may be placed if the Quantiferon TB gold test is indeterminate. Patients must have a negative Quantiferon TB Gold (or tuberculin skin test) or evidence of appropriate treatment prior to study entry.

1.8 Patients must be able to understand and sign a written informed consent document and complete study-related procedures and questionnaires.

EXCLUSION CRITERIA

2.1 Enrollment in any other investigational treatment study or use of an investigational agent, or has not yet completed at least 3 half-lives since ending another investigational device or drug trial.

2.2 History of treatment with canakinumab within the 12 months prior to study initiation.

2.3 History of anakinra use.

2.4 History of phototherapy within 2 weeks prior to study initiation.

2.5 Patients may NOT concurrently be on biologic therapy such as etanercept, adalimumab, alefacept, infliximab, rituximab or rilonacept. If there is a history of use of biologic agents, there must be a washout period of at least 3 half-lives prior to study initiation.

2.6 Subjects who experience a significant flare after discontinuation of a tumor necrosis factor (TNF) inhibitor as part of this study that requires urgent medical management or hospitalization, or in the estimation of the principal investigator poses excessive risk to the patient to enter the study.

2.7 Other defined dermatologic conditions which may include pustules as part of the clinical presentation, but which clinically and/or histologically do not resemble pustular psoriasis. Examples include, but are not limited to acute generalized exanthematous pustulosis (Acute generalized exanthematous pustulosis (AGEP), a drug-induced pustular dermatosis typically caused by beta-lactam antibiotics, tetracyclines, oral antifungals and other drugs), bacterial or fungal folliculitis, cutaneous candidiasis, tinea pedis, tinea corporis, neutrophilic eccrine hidradenitis or eosinophilic pustular folliculitis (Ofuji syndrome).

2.8 Known diagnosis of Deficiency of the interleukin-1 receptor antagonist (DIRA).

2.9 History of allergic reactions attributed to compounds of similar chemical or biologic composition to anakinra or other agents used in study. Known hypersensitivity to Chinese hamster ovary (CHO)-cell derived biologics or any components of anakinra.

2.10 Treatment with a live virus vaccine during the 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study.

2.11 Patients with active or untreated malignancy-- with the exception of cutaneous basal or squamous cell carcinomas, or in situ cervical carcinoma-- are ineligible because of the immunomodulating effects of anakinra. The risk of recurrent malignancy secondary to this drug is unknown.

2.12 Presence of active infection. History of exposure to TB (positive purified protein derivative (PPD) or Quantiferon TB gold) who have not been treated with a TB prophylaxis regimen for at least one month.

2.13 Chest x-ray demonstrating pleural scarring and/or calcified granuloma consistent with prior or current untreated TB.

2.14 History of chronic or recurrent infection including but not limited to human immunodeficiency virus (HIV), hepatitis B or hepatitis C.

2.15 Individuals with severe or uncontrolled recurrent cutaneous infections who are considered at elevated risk for serious infection on anakinra therapy will be excluded per physician discretion.

2.16 Presence of other known significant autoimmune or inflammatory disease. Examples include major chronic infectious/inflammatory/immunologic diseases such as systemic lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome and periodic fever syndromes.

2.17 Other immunoregulatory or immunodeficiency diseases, such as multiple sclerosis.

2.18 Individuals with life-threatening or disabling inflammation of the eyes, gut or joints requiring urgent or immediate medical attention, or at the physicians discretion.

2.19 Subjects for whom there is concern about compliance with the protocol procedures.

2.20 Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled or unmonitored psychiatric illness/social situations, or history of congestive heart failure, unstable angina pectoris or medically significant cardiac arrhythmia that would limit compliance with study requirements.

2.21 Presence of other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject enrollment inappropriate.

2.22 The effects of anakinra on the developing human fetus are unknown. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Females of childbearing potential must have a negative serum pregnancy test at screening. Females must also have a negative serum pregnancy test at baseline and prior to performance of any radiologic procedure or administration of study medication and during each National Institutes of Health (NIH) visit. Lactating mothers will discontinue breastfeeding prior to study enrollment.

2.23 Pregnant or lactating females. Women of non-childbearing potential is defined as women who are postmenopausal (no menses for > one year) or who have had a hysterectomy and will not require Beta-Human Chorionic Gonadotropin (B-HCG) testing

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Cowen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-AR-0071.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Week 4 Level 1 Only: Anakinra Week 4 Level 1, 100mg administered subcutaneously daily.
- Week 4 Level 1 Followed by Week 8 Level 2: Anakinra Week 4 Level 1, 100mg administered subcutaneously daily followed by Week 8 Level 2, 200 mg.
- Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2: Anakinra Week 4 Level 1, 100mg administered subcutaneously daily followed by Week 8 Level 2, 200 mg, followed by Week 12 Level 2, 200mg.
- Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3: Anakinra Week 4 Level 1, 100mg administered subcutaneously daily followed by Week 8 Level 2, 200 mg, followed by Week 12 Level 3, 300mg (participants 75kg only).
Period: Overall Study
Arm/Group | Week 4 Level 1 Only | Week 4 Level 1 Followed by Week 8 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3
Started | 1 | 3 | 2 | 12
Completed | 0 | 0 | 2 | 12
Not Completed | 1 | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Participant noncompliance | 0 | 1 | 0 | 0
Not completed — Refused further treatment | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Week 4 Level 1 Only | Week 4 Level 1 Followed by Week 8 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3 | Total
Number analyzed (Participants) | 1 | 3 | 2 | 12 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 2 | 11 | 17
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (0) | 45.43 (1.51) | 49.9 (20.51) | 51.55 (11.53) | 50.21 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 11 | 15
  Male | 1 | 1 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 3 | 1 | 12 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 1 | 2 | 1 | 8 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Treated With Anakinra Who Achieve 50% Disease Improvement by the End of Week 12, as Measured by Total Body Surface Area Involvement (TBSAI50)
Description: Total Body Surface Area Involvement (TBSAI) is defined as the amount of total amount of active disease involvement on a given patient. 50% improvement was the amount of change that we judged at the start of the study would qualify as significant improvement.
Time Frame: 12 Weeks
Population: 14/18 were analyzed because 4 pts did not meet the study primary endpoint (stayed on treatment until 12 wks). The study was not powered nor intended to study/compare differences between dose levels. The dose escalation was done for safety purposes rather than dose finding.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: All participants that received Anakinra 100mg, 200mg, and 300mg administered subcutaneously daily for 12 weeks.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Participants | 7

2. Other Pre Specified Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Up to 16 weeks for participants who completed active treatment (12 weeks) and 4 weeks of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Week 4 Level 1 Only | Week 4 Level 1 Followed by Week 8 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3
Number analyzed (Participants) | 1 | 3 | 2 | 12
Participants | 1 | 3 | 2 | 12

3. Other Pre Specified Outcome: Average Change in Total Body Surface Area Index (TBSAI)
Description: Median difference in affected area of plaque and pustular disease between baseline and week 12.
Time Frame: Baseline and 12 Weeks
Population: The study was not powered nor intended to study/compare differences between dose levels. The dose escalation was done for safety purposes rather than dose finding.
Measure: Median (Inter-Quartile Range); unit: Percentage of total skin involvement
Arm/Group | All Participants
Number analyzed (Participants) | 14
Percentage of total skin involvement | -0.9 [-1.8 to 0.0]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.033, Wilcoxon Signed Rank Test

ADVERSE EVENTS:
Time Frame: Up to 16 weeks for participants who completed active treatment (12 weeks) and 4 weeks of follow-up.
Arm/Group | Week 4 Level 1 Only | Week 4 Level 1 Followed by Week 8 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/2 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/3 | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 2/2 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Week 4 Level 1 Only (N=1) | Week 4 Level 1 Followed by Week 8 Level 2 (N=3) | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 (N=2) | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3 (N=12)
Skin and subcutaneous tissue disorders - Other, Flare of Pustular Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Week 4 Level 1 Only (N=1) | Week 4 Level 1 Followed by Week 8 Level 2 (N=3) | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 2 (N=2) | Week 4 Level 1, Followed by Week 8 Level 2, Followed by Week 12 Level 3 (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
GGT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (4) | 0 (0) | 7 (31)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations - Other, L foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (3) | 2 (2) | 9 (10)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (4) | 6 (9)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (8)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (8)
Respiratory, thoracic and mediastinal disorders - Other, Running Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Eye disorders - Other, (Stye L eye) (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Eye disorders - Other, (Stye R eye) (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Hiradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT01794117/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT01794117/ICF_001.pdf